CLINICAL TRIAL: NCT00835822
Title: Multicenter, Prospective, Randomized, Double-Blind Study to Assess the Therapeutic Efficacy and Safety of the Use of Venocur Triplex® in Patients With Chronic Venous Insufficiency
Brief Title: Efficacy and Safety of the Use of Venocur Triplex® in Patients With Chronic Venous Insufficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Statistika Consultoria Ltda (Industry)
Responsible Party: Suely Kumagai Inoue, Abbott Laboratórios do Brasil Ltda.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRAZ-03-003
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Venous Insufficiency
Keywords: Chronic Venous Insufficiency, Venocur Triplex®
MeSH Terms: conditions — Venous Insufficiency | interventions — phenopyrazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Arm treated with Investigational product.
  Interventions: Drug: Venocur Triplex®
- B (Placebo Comparator): Arm treated with placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Venocur Triplex® — Administered by oral route, two coated tablets per day, after the meals (breakfast and dinner), with some liquid, but not with alcoholic beverages.
  Other Names: ABT-401; venopyronum; Venocur Triplex
  Arms: A
Drug: placebo — Administered by oral route, two coated tablets per day, after the meals (breakfast and dinner), with some liquid, but not with alcoholic beverages.
  Arms: B

SUMMARY:
The purpose of this study is to assess the therapeutic efficacy and safety of Venocur Triplex®, administered BID for 60 days in patients with Chronic Venous Insufficiency rated between CEAP 2 and 4, in comparison to a Placebo group.

ELIGIBILITY:
Inclusion Criteria:

* The patient has confirmed his/her willingness to participate in the study, after being informed about all the aspects of the study that might be relevant for his/her decision to participate, and has signed and dated the informed consent form, as approved by the Institutional Review Board/ Ethics Committee (IRB/EC)
* Patients of both sexes, aged above 18 years and below 65 years
* Presence of uni- or bilateral varicose veins with CVI, in both sexes
* The patient's CVI is rated between functional classes CEAP 2 and 4
* Present at least one symptom of CVI prior to the study - leg pains, cramps, fatigue, heavy legs sensation.

Exclusion Criteria:

* If female, the patient has circulatory disorders exclusively during the pre-menstrual period
* If the patient is pregnant or breastfeeding
* The patient has received anticoagulants less than 15 days before study start
* The patient has used steroids or anti-inflammatory drugs less than 8 days before study start
* The patient has received radio or chemotherapy less than 7 days before study start
* The patient has used diuretics, phlebotrophic and venoactive drugs over the past 8 days before enrollment in the study
* The patient has used compression stockings less than 8 days before study start
* Trauma or surgical treatment over the past 30 days before study start
* Prior surgical treatment related to CVI (past 12 months for surgery and past 6 months for sclerotherapy)
* Immobilization of lower limbs over the past 6 months
* Known allergy to the product's ingredients
* Presence of chronic inflammatory diseases (rheumatoid arthritis, for instance), severe chronic infectious diseases (AIDS, tuberculosis, hanseniasis, etc.)
* The patient has suffered from phlebitis or deep venous thrombosis in the past 6 months before the study
* Fibrous lymphedema, primary or secondary lymphedema and lipoedema;
* Concomitant erysipelas
* Active fungal infections of the lower limbs
* Peripheral arteries disease, cerebrovascular or coronary disease
* Severe systemic conditions (heart failure, liver, pulmonary or kidney failure, active neoplastic disease, severe arterial hypertension, uncontrolled diabetes, among others), over the past 6 months before study start
* Hematocrit: < 32.0 mL RBC/dL for women and < 36.0 mL RBC/dL for men
* Hemoglobin: < 11.0 mL g/dL for women and < 12.0 mL g/dL for men;
* Total protein and fractions: Total protein < 6.4 g/dL, Albumin < 4.0 g/dL, Globulin < 1g/dL and Albumin/Globulin < 0.9%
* Serum creatinine: > 1.0 mg/dL for women and > 1.2 mg/dL for men or if patient in dialysis
* Aminotranferases (SGOT/AST and/or SGPT/ALT) more than twice the upper normal limit
* Participation in study with similar objectives over the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2005-05; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Reduction of the score of the CVI symptoms, based on symptoms as leg pains, cramps, fatigue, aching legs, heavy legs sensation, heat or burning sensation and paresthesia (tingling/numbness) | 60 days
Improvement of each CVI symptoms - leg pains, cramps, fatigue, aching legs, heavy legs sensation, heat or burning sensation and paresthesia (tingling/numbness);
Safety Assessment through the adverse events reports

SECONDARY OUTCOMES:
Reduction of edema in patients rated between CEAP 3 and 4, as compared to the Placebo group
Effects of the study drug on the patient's quality of life using questionnaires SF-36 and CVIQ | 60 days
The global clinical improvement of the patient with CVI, using the CGI (Clinical Global Impression) scale. | 60 days

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Belo Horizonte, Minas Gerais
  - Botucatu, São Paulo
  - Marília, São Paulo
  - São Paulo, São Paulo